CLINICAL TRIAL: NCT06952738
Title: Investigating Periprosthetic Fracture Culture Positivity in Patients With Hip and Knee Arthroplasties
Brief Title: Investigating Periprosthetic Fracture Cultures in Arthroplasty
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB25-0498
Record Dates: First submitted 2025-04-23; First posted 2025-05-01 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Periprosthetic Fracture Around Prosthetic Joint Implant
Keywords: Periprosthetic fractures; synovial fluid; prosthetic joint infections
MeSH Terms: conditions — Periprosthetic Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will be collecting synovial fluid and tissue cultures from hips and knees with periprosthetic fractures and will be monitoring the cultures for 14 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Periprosthetic Fractures: This group will be all patients enrolled in the study: they will all have periprosthetic hip or knee fractures.
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — The investigators are only looking to see the rate of positivity of the cultures as well as what the organisms that are found in the cultures are.

SUMMARY:
This study aims to improve how doctors diagnose infections in patients with broken bones around joint replacements. Currently, there are no clear guidelines to help determine when an infection is present, making treatment decisions difficult. By studying how often infections are found through lab tests and identifying factors that predict infection, the investigators hope to create better ways to diagnose and care for these patients.

DETAILED DESCRIPTION:
All steps in the protocol will be completed under the standard of care for our hospital's orthopedic joints and trauma surgeons. All patients identified under the inclusion criteria will undergo preoperative imaging. In accordance with current standards of care, patients with periprosthetic fractures (PPFs) around the hip will receive three views of X-rays of the hip and femur as well as the anterior-posterior view of the pelvis. Likewise, patients with PPFs around the knee will undergo X-rays that include the knee and femur. No advanced imaging (Computed Tomography, Magnetic Resonance Imaging, etc.) will be obtained for the purpose of this study.

Preoperative laboratory analysis will include C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR) as inflammatory markers. Intraoperative synovial fluid analysis will be performed using synovial white blood cell (WBC) count and polymorphonuclear (PMN) percentage. Three cultures will be obtained from the involved joint fluid and tissue, and incubated for 14 days for analysis of aerobic, anaerobic bacterial cultures, fungal and acid-fast bacilli (AFB) analysis. The cultures will be collected from synovial fluid, peri-implant femoral synovium/periosteum, peri-implant tibial or acetabular synovium/periosteum. These laboratory tests and cultures are part of the standard protocol our surgeons have determined for their patient care.

Based on the Musculoskeletal Infection Society (MSIS) criteria for positive histology intraoperative histology will be performed utilizing frozen section analysis. These slides will be isolated from synovium, peri-implant femoral synovium/periosteum, and peri-implant tibial or acetabular synovium/periosteum. Additional cultures may be sent at discretion of surgeon but would not be included in analysis.

Per institutional protocol, preoperative cefazolin and vancomycin will be administered intravenously and continued for 24 hours perioperatively. Patients who are allergic to vancomycin will receive daptomycin, and those who are allergic to beta-lactam drugs including cephalosporins will be given gentamicin. No intra-articular antibiotics will be routinely administered.

All cultures will be followed until final. If cultures become positive, our institutional infectious disease (ID) department will be consulted for further recommendations and consideration for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old) with periprosthetic fractures around primary or revision hip or knee arthroplasty
* Patients requiring operative management for these fractures (fixation or revision arthroplasty)
* Patients presenting to the University of Chicago Medical Center during two (2) year period (October 2025 to October 2027)

Exclusion Criteria:

* Patients undergoing non-operative management for periprosthetic fractures
* Any documented or reported history of past prosthetic joint infection of the involved joint
* Sinus tract at the time of presentation at the involved joint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This population would include all consenting patients older than 18 years who present to the University of Chicago Medical Center with periprosthetic hip or knee fractures and will require operative management of the fracture or infection.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Culture Positivity Rates | From enrollment to the end of treatment at 14 days.
  This outcome measure is the percentage of cultures that grow organisms among the population

SECONDARY OUTCOMES:
Rate of Complications | From date of surgery to one year after the specific participant's surgery.
  Number of participants with surgery-related complications within one year after their surgeries.
Culture Organisms | From surgery date to 14 days after surgery.
  The names, number, and frequency of organisms being found in the cultures.
Treatments Used | From enrollment to one year after surgery.
  The list of antibiotics used for treating organisms found to be positive in the cultures.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Wallace, MD, Principal Investigator — The University of Chicago Department of Orthopaedic Surgery
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parvizi J, Tan TL, Goswami K, Higuera C, Della Valle C, Chen AF, Shohat N. The 2018 Definition of Periprosthetic Hip and Knee Infection: An Evidence-Based and Validated Criteria. J Arthroplasty. 2018 May;33(5):1309-1314.e2. doi: 10.1016/j.arth.2018.02.078. Epub 2018 Feb 26. PMID 29551303
- [Background] McArthur BA, Abdel MP, Taunton MJ, Osmon DR, Hanssen AD. Seronegative infections in hip and knee arthroplasty: periprosthetic infections with normal erythrocyte sedimentation rate and C-reactive protein level. Bone Joint J. 2015 Jul;97-B(7):939-44. doi: 10.1302/0301-620X.97B7.35500. PMID 26130349
- [Background] Schinsky MF, Della Valle CJ, Sporer SM, Paprosky WG. Perioperative testing for joint infection in patients undergoing revision total hip arthroplasty. J Bone Joint Surg Am. 2008 Sep;90(9):1869-75. doi: 10.2106/JBJS.G.01255. PMID 18762646
- [Background] Shah RP, Plummer DR, Moric M, Sporer SM, Levine BR, Della Valle CJ. Diagnosing Infection in the Setting of Periprosthetic Fractures. J Arthroplasty. 2016 Sep;31(9 Suppl):140-3. doi: 10.1016/j.arth.2015.08.045. Epub 2016 Mar 17. PMID 27067465
- [Background] Preston S, Somerville L, Lanting B, Howard J. Are Nucleated Cell Counts Useful in the Diagnosis of Infection in Periprosthetic Fracture? Clin Orthop Relat Res. 2015 Jul;473(7):2238-43. doi: 10.1007/s11999-015-4162-8. PMID 25631172
- [Background] Chevillotte CJ, Ali MH, Trousdale RT, Larson DR, Gullerud RE, Berry DJ. Inflammatory laboratory markers in periprosthetic hip fractures. J Arthroplasty. 2009 Aug;24(5):722-7. doi: 10.1016/j.arth.2008.05.026. Epub 2008 Sep 11. PMID 18789633
- [Background] Austin MS, Ghanem E, Joshi A, Lindsay A, Parvizi J. A simple, cost-effective screening protocol to rule out periprosthetic infection. J Arthroplasty. 2008 Jan;23(1):65-8. doi: 10.1016/j.arth.2007.09.005. PMID 18165031
- [Background] van den Kieboom J, Tirumala V, Xiong L, Klemt C, Kwon YM. Concomitant Hip and Knee Periprosthetic Joint Infection in Periprosthetic Fracture: Diagnostic Utility of Serum and Synovial Fluid Markers. J Arthroplasty. 2021 Feb;36(2):722-727. doi: 10.1016/j.arth.2020.08.029. Epub 2020 Aug 18. PMID 32893059
- [Background] Barberis L, Abdelrahman T, Driscoll DA, Dasci MF, Gehrke T, Citak M. Unexpected Positive Cultures in Hip and Knee Periprosthetic Fractures. J Arthroplasty. 2024 Jul;39(7):1834-1839. doi: 10.1016/j.arth.2024.01.030. Epub 2024 Jan 18. PMID 38244640
- [Background] Shichman I, Roof M, Askew N, Nherera L, Rozell JC, Seyler TM, Schwarzkopf R. Projections and Epidemiology of Primary Hip and Knee Arthroplasty in Medicare Patients to 2040-2060. JB JS Open Access. 2023 Feb 28;8(1):e22.00112. doi: 10.2106/JBJS.OA.22.00112. eCollection 2023 Jan-Mar. PMID 36864906
- [Background] Sloan M, Premkumar A, Sheth NP. Projected Volume of Primary Total Joint Arthroplasty in the U.S., 2014 to 2030. J Bone Joint Surg Am. 2018 Sep 5;100(17):1455-1460. doi: 10.2106/JBJS.17.01617. PMID 30180053